CLINICAL TRIAL: NCT00048308
Title: Effect of Pexelizumab on All-Cause Mortality and Myocardial Infarction in Patients Undergoing Coronary Artery Bypass Graft Surgery With Cardio-Pulmonary Bypass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000099; PRIMO-CABG
Record Dates: First submitted 2002-10-29; First posted 2002-10-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cardio-pulmonary Bypass; Coronary Artery Bypass Graft
Keywords: CABG
MeSH Terms: interventions — pexelizumab

INTERVENTIONS:
Drug: pexelizumab

SUMMARY:
During a heart bypass procedure, a substance called "complement" is released by the body. This complement causes inflammation, which can lead to side effects such as chest pain, heart attacks, heart failure, or impairment of memory, language and motor skills. The purpose of this study is to find out if the study drug (pexelizumab), which blocks complement release, can reduce such side effects and be taken safely.

ELIGIBILITY:
INCLUSION CRITERIA:

The study population will be drawn from patients undergoing CABG or CABG plus valve surgery using a bypass pump. In addition, they must meet all of the following criteria:

* be at least 18 years of age;
* have one or more of the following risk factors:
* diabetes mellitus;
* prior CABG;
* the need for urgent intervention, defined according to the American College of Cardiology/ American Heart Association (ACC/AHA) guidelines as being patients who are required to stay in the hospital, but may be scheduled and operated on within a normal scheduling routine, excluding patients who have had a MI within 48 hours of CABG;
* female;
* history of a neurologic event (cerebrovascular accident, transient ischemic attack or carotid endarterectomy);
* history of congestive heart failure (New York Heart Association [NYHA]Class III or IV);
* history of 2 myocardial infarctions, or a myocardial infarction that occurred greater than 48 hours but less than four (4) weeks prior to CABG;
* provide Informed Consent.

EXCLUSION CRITERIA:

A patient will be ineligible for study entry if he/she meets any of the following exclusion criteria:

* has planned aortic dissection repair and/or requires aortic root reconstruction;
* requires salvage intervention as defined by the ACC/AHA guidelines as being ongoing cardiopulmonary resuscitation on the way to the operating room;
* has current cardiogenic shock, acute left ventricular rupture, acute septal rupture or acute papillary muscle rupture;
* has uncontrolled diabetes, defined as a documented plasma blood glucose value > 400 mg/dl (22.2 mmol/L) within three (3) days before surgery;
* has a history of renal failure and a serum creatinine value greater than 3.0 mg/dl;
* has a history of chronic hepatic failure and/or hepatic cirrhosis;
* has a history of malignancy, excepting basal cell carcinoma and malignancies in remission (greater than 2 years);
* has any active bacterial or other infection which is clinically significant, in the opinion of the investigator (e.g. evaluate the evidence based on WBC, temperature, cultures, etc. as appropriate for the patient);
* has any serious medical condition which, in the opinion of the investigator is likely to alter the patient's course of recovery or the evaluation of the study medication's safety;
* has a history of alcohol or drug abuse within the past year;
* has a known or suspected hereditary complement deficiency;
* has participated in any other investigational drug study or was exposed to an investigational agent or device within 30 days of randomization;
* is receiving, or is planning to receive, any other investigational drug or device, or will participate in any other research study during the trial;
* is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2002-01 (Actual); Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (185):
- United States (167):
  - Baptist Medical Center Cardiology, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - IMC-Diagnostic and Medical Clinic, Mobile, Alabama
  - Desert Samaritan - Lutheran Heart, Mesa, Arizona
  - Good Samaritan Regional Medical Center, Phoenix, Arizona
  - Saguaro Clinical Research, Tucson, Arizona
  - Southern Arizona VAMC, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - University of Arkansas, Little Rock, Arkansas
  - Brotman Medical Center, Beverly Hills, California
  - Cardiovascular Associates of the Peninsula, Burlingame, California
  - Seton Medical Center, Daly City, California
  - St. Jude Medical Center, Fullerton, California
  - Apex Cardiology, Inglewood, California
  - Huntington Memorial Hospital, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - St. Vincent's Hospital, Los Angeles, California
  - University of California - Los Angeles, Los Angeles, California
  - Crozer-Chester Medical Center, Oakland, California
  - Tri-City Medical Center, Oceanside, California
  - Mercy General Hospital, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - Kaiser Foundation Hospital, San Francisco, California
  - UCSF Moffitt-Long Hospital, San Francisco, California
  - South Denver Cardiology Associates, Denver, Colorado
  - Western Cardiology Associates, Denver, Colorado
  - Heart and Vascular Clinic of Northern CO, Fort Collins, Colorado
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Cardiology Associates, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - VA Medical Center - Washington DC, Washington D.C., District of Columbia
  - Florida Cardiovascular Research, Atlantis, Florida
  - Morton Plan Mease Health Care, Clearwater, Florida
  - Heart Group Research, Fort Lauderdale, Florida
  - Gulf Bay Cardiovascular and Thoracic Associates, Hudson, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Brevard Cardiology Group, PA, Merritt Island, Florida
  - Medical Research Unlimited, Miami, Florida
  - Florida Heart Institute at Florida Hospital, Orlando, Florida
  - Orlando Heart Center, Orlando, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Ford Research Center, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northside Hospital ans Heart Institute, St. Petersburg, Florida
  - Tallahassee Memorial Regional Medical Center, Tallahassee, Florida
  - Pepin Heart and Vascular Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - University Hospital, Augusta, Georgia
  - VA Medical Center- Atlanta, Decatur, Georgia
  - VA Medical Center - Dubin, Macon, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Medical Center, Honolulu, Hawaii
  - Northwestern Univ. Medical Center, Chicago, Illinois
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Illinois - Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare Evanston Hospital, Evanston, Illinois
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - Community Hospital, Indianapolis, Indiana
  - St. Vincent's Medical Center, Indianapolis, Indiana
  - Iowa Heart Center - Laurel, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - University of Kansas City Medical Center, Kansas City, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Turuo Infirmary, New Orleans, Louisiana
  - Methodist Hospital, New Orleans, Louisiana
  - Alton Ochsner Medical Foundation - Brent House, New Orleans, Louisiana
  - Cardiac Centers of Louisiana, Shreveport, Louisiana
  - Cardiovascular Institute of the South, Thibodaux, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Midatlantic Cardiovascular Associates, Towson, Maryland
  - St. Joseph's Hospital, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Thoracic and Cardiovascular Institute, Lansing, Michigan
  - West Shore Cardiology Research Department, Muskegon, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - St. Luke's Hospital-Duluth, Duluth, Minnesota
  - St. Mary's Duluth Health System, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Medical Center, Minneapolis, Minnesota
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Park Nicollet Health Research Center, Saint Louis Park, Minnesota
  - Mississippi Center for Clinical Research, Jackson, Mississippi
  - Cardiology diagnostics, Ltd., City of Saint Peters, Missouri
  - St. Luke's Hospital - Mid-America Heart Institute, Kansas City, Missouri
  - Christian North East Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Garden State Cardiology, Paramus, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - United Health Services, Johnson City, New York
  - New York Presbyterian Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Albert Einstein Hospital, The Bronx, New York
  - Westchester County Medical Center, Valhalla, New York
  - Asheville Cardiothoracic Surgeons, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - West forest School of Medicine, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Summa Health Systems, Akron, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - Good Samaritan Hospital -Seton Center, Cincinnati, Ohio
  - Tri Health Bethesda North Hospital, Cincinnati, Ohio
  - University Hopital of Cleveland, Cleveland, Ohio
  - Mt. Carmel West, Columbus, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - North Ohio Heart Center, Sandusky, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Northwest Surgical Associates, Portland, Oregon
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - The Heart Center, Doylestown, Pennsylvania
  - North Memorial Pain Institute, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Chester County Cardiovascular Center, West Chester, Pennsylvania
  - The Chattanooga Heart Institute Cardiovascular Group, P.C., Chattanooga, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Parkway Cardiovascular Associates, Oak Ridge, Tennessee
  - Brackenridge Hospital, Austin, Texas
  - Seton Medical Center, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - VA Medical Center - Houston, Houston, Texas
  - Texas Tech University Health Center, Lubbock, Texas
  - South Texas Cardiovascular Consultants Clinical Research Center, San Antonio, Texas
  - South Texas VA Health Care, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cardiovascular and Thoracic Surgery Associates, Arlington, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carillion Roanoke Hospital, Roanoke, Virginia
  - VA-Medical Center -Seattle Cardiology, Seattle, Washington
  - University of Washington, Seattle, Washington
  - FHS Research Center, Tacoma, Washington
  - Tacoma General Hospital, Tacoma, Washington
  - Camcare Health Education & Research Institute, Charleston, West Virginia
  - Appleton Medical Center, Appleton, Wisconsin
  - Gundersen-Lutheran Hospital, La Crosse, Wisconsin
  - Wisconsin Center for Clinical Research, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cardiovascular Research and Education Foundation, Inc., Wausau, Wisconsin
- Canada (18):
  - Makenzie Health Science Center, Edmonton, Alberta
  - Cathy Metcalfe Research Consultants, Delta, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute, Victoria, British Columbia
  - University of Manitoba Health Science Centre, Winnipeg, Manitoba
  - Health Science Centre, Winnipeg, Manitoba
  - New Brunswick Heart Center, Saint John, New Brunswick
  - General Hospital Health Science Center, St. John's, Newfoundland and Labrador
  - Dalhousie University, Halifax, Nova Scotia
  - McMaster Clinic, Hamilton, Ontario
  - Sunnybrook & Women's College Health Science Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - University of Montreal, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Hopital Laval, Québec, Quebec
  - Regina General Hospital, Regina, Saskatchewan